CLINICAL TRIAL: NCT00238667
Title: Cervical Artery Dissection in Stroke Study
Brief Title: To Determine the Feasibility of a Clinical Trial Comparing Anticoagulants Versus Antiplatelets in the Acute Treatment of Patients With Cervical Artery Dissection
Acronym: CADISS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: The Stroke Association, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAMER5UA; 2006-002827-18 (EudraCT Number); 04.0287 (Other: Sponsor St Georges University of London); 04/Q0803/15 (Other: REC/IRB reference); 04/Q0803/215 (Other: REC/IRB reference); TSA2004/16
Record Dates: First submitted 2005-10-11; First posted 2005-10-13 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2005-09

CONDITIONS: Cervical Artery Dissection; Carotid Artery Dissection; Vertebral Artery Dissection; Stroke
Keywords: Extracranial carotid artery dissection; Dissection and stroke
MeSH Terms: conditions — Vertebral Artery Dissection; Stroke | interventions — Aspirin; Dipyridamole; Clopidogrel; Anticoagulants; Heparin; Dalteparin; Warfarin

ARMS (2):
- Anti-platelet therapy (Active Comparator): Aspirin, Dipyridamole, clopidogrel alone or in dual therapy
  Interventions: Drug: Antiplatelet (Aspirin, Dipyridamole, clopidogrel)
- Anti-coagulant (Active Comparator): Warfarin, unfractionated heparin, enoxaparin, dalteparin, tinzaparin aiming for an INR in range of 2-3. Local protocols for Heparin can be used
  Interventions: Drug: Anticoagulant (Unfractionated Heparin, LMW Heparin, Warfarin)

INTERVENTIONS:
Drug: Antiplatelet (Aspirin, Dipyridamole, clopidogrel)
  Other Names: Aspirin, Dipyridamole, clopidogrel
  Arms: Anti-platelet therapy
Drug: Anticoagulant (Unfractionated Heparin, LMW Heparin, Warfarin)
  Other Names: Unfractionated Heparin, LMW Heparin, Warfarin
  Arms: Anti-coagulant

SUMMARY:
This is a feasibility study to determine if a sufficient number of patients can be recruited throughout the United Kingdom and whether sufficient endpoints can be generated for a full scale therapeutic trial of anticoagulants versus antiplatelets in acute cervical artery dissection treatment.

DETAILED DESCRIPTION:
ST. GEORGE'S HEADED NOTEPAPER

CADISS FEASIBILITY STUDY (Cervical Artery Dissection in Stroke Study) PROTOCOL

Aim:

To determine the feasibility of a clinical trial comparing antiplatelet therapy with anticoagulation in the acute treatment of patients with cervical artery dissection. Specifically to address whether:

1. There are sufficient clinical endpoints to provide the power to determine treatment effect;
2. Adequate numbers of patients can be recruited.

Dissection of the carotid and vertebral arteries is a major cause of stroke in persons < 50 years of age, mainly due to embolism from clot sealing the tear. At present physicians treat these patients with anticoagulants or antiplatelet drugs to prevent further stroke, but neither therapy is evidence-based. Anticoagulants may be powerful anti-embolic agents but are also more dangerous than aspirin, and potentially could encourage further dissection. Most published studies are flawed by retrospective data, with no reference to the number of patients in the original study cohort and do not include the critical principles of randomisation and 'blinding'.

Proposal of present 'feasibility'study:

The only prospective data available (1) suggest that anticoagulants are more effective than antiplatelet agents in reducing further TIA and stroke after dissection, but the numbers were small and lack reliable statistical confirmation. This study was not a randomised controlled trial and therefore may be open to bias in selection of treatment. As well, it found that most recurrent events occur within the first month and thereafter the number tails off. A total of about 1800 patients for a two armed therapeutical trial was necessary to be calculated on these data.

Authors of a previous Cochrane review (2) reviewing available published literature calculated that a total of about 2000 patients (1000 in each treatment arm) is needed for a blinded randomised trial of anticoagulants versus antiplatelet agents. This would need a major, probably international, study involving over 50 centres, and would be an expensive undertaking. Prior to starting such a study it is important to determine whether this would be feasible. This is particularly important for carotid and vertebral dissection which is a frequently missed diagnosis, at least during the acute phase. Limited natural history outcome data suggest the risk of recurrent stroke and TIA following carotid and vertebral dissection is only markedly raised during the first week to month (1, 3) and therefore early identification and recruitment of patients are essential if any treatment effect is to be demonstrated.

For these reasons, a feasibility study is essential before any large scale clinical trial. Specifically, two things need to be determined. Firstly, whether a sufficient number of patients can be recruited sufficiently early from participating centres. Secondly, in view of the limited data on the rate of recurrent TIA and stroke in patients with recent dissection, we need more data to obtain a robust estimate of early risk to inform power calculations for a large scale study.

A preliminary informal survey conducted by Clinical Neurosciences, St. George's University of London, in association with the Association of British Neurologists, has indicated that at least 27 neurologists/stroke physicians throughout the UK would be interested in collaborating and enrolling consecutive consenting patients into such a study comparing anticoagulation or antiplatelet therapy.

Methods:

This will be a randomised multicentre single blind study comparing antiplatelet therapy with anticoagulation for patients with carotid and vertebral dissection. Recruitment must be within seven days of onset of symptoms.

Inclusion Criteria:

1. Extracranial carotid or vertebral artery dissection with symptom onset within the last 7 days. This includes:

   1. Ipsilateral TIA or stroke
   2. Ipsilateral Horner's syndrome or neck pain with known date of onset
2. Imaging evidence of definite or probable dissection on magnetic resonance imaging (MRI)/magnetic resonance angiography (MRA), computed tomography angiography (CTA) or ultrasound (patients can be initially randomised on ultrasound alone but subsequent MR or CTA confirmation is needed)

Exclusion Criteria:

1. Intracranial cerebral artery dissection
2. Symptom onset after 7 days
3. Contraindications to either antiplatelet agents or anticoagulation therapy
4. Patient refusal to consent
5. Patients who are undergoing angioplasty and stenting or surgery for treatment of their dissection

Treatment:

Patients will be randomised to either antiplatelet or anticoagulation therapy allocated on a single blind basis and continued for six months.

1. Antiplatelet therapy: Aspirin 75-300 mg daily, aspirin and dipyridamole or clopidogrel alone
2. Anticoagulation with heparin (either unfractionated heparin or a therapeutic dose of low molecular weight heparin) followed by warfarin aiming for an INR in the range 2.5-4. Local protocols for heparin therapy can be used.

Primary Endpoint:

Ipsilateral stroke, transient ischaemic attack or vascular death within 6 months from randomisation

Secondary Endpoint:

1. TIA and stroke in other cerebral vascular territories
2. Recanalisation on repeat imaging at 6 months.

Imaging Protocol:

The diagnosis of dissection is based on different modalities in different centres. Centres should use their usual imaging protocol to diagnose dissection. Diagnosis on the basis of MRI with cross-sectional imaging through the artery wall, MRA, CT angiography, intra-arterial angiography, and ultrasound (later confirmed by MR or CTA) are all acceptable.

Patients can be randomised if the HQ radiologist (Dr. Clifton) agrees that the diagnosis is probable or definite. Hard copies of imaging must be recorded for central reading.

The primary analysis will include only those patients judged to have probable or definite dissection on central reading of the hard copies.

Randomisation:

Randomisation will be via 24 hour randomisation service provided by the University of Aberdeen Health Services Research Unit.

The local investigator will personally contact this service at 0800 387 4444 and the Centre will give the investigator a code number, known only to the randomisation centre and local investigator.

Trial Management:

The study will be coordinated from Clinical Neuroscience at St. George's, University of London. The principal co-investigators are Professor John Norris and Professor Hugh Markus. The principal neuroradiological investigator, responsible for assessment of hard copies of imaging, is Dr Andrew Clifton. The trial will be coordinated by a clinical fellow funded by a project grant from The Stroke Association.

References

1. Beletsky V, Nadareishvili Z, Lynch J, Shuaib A, Woolfenden A, Norris JW; Canadian Stroke Consortium (2003) Cervical Arterial Dissection; Time for a Therapeutic Trial? Stroke Dec; 34(12)2856-60
2. Lyrer P, Engelter S. Antithrombotic drugs for carotid artery dissection. Cochrane Review Oxford,UK. Cochrane Library 2002. Issue 1
3. Biousse V, D'Anglejan-Chatillon J, Touboul PJ, Amarenco P, Bousser MG (1995) Timecourse of Symptoms in Extracranial Carotid Artery Dissections. A Series of 80 patients Stroke Feb; 26(2)

ELIGIBILITY:
Inclusion Criteria:

1. Extracranial carotid or vertebral artery dissection with symptom onset within the last 7 days. This includes:

   1. Ipsilateral transient ischemic attack or stroke
   2. Ipsilateral Horner's syndrome or neck pain with known date of onset.
2. Imaging evidence of definite or probable dissection on MRI/MRA, CTA or ultrasound.

Exclusion Criteria:

1. Intracranial cerebral artery dissection
2. Symptom onset after 7 days
3. Contraindication to either antiplatelet agents or anticoagulation therapy
4. Patient's refusal to consent
5. Patients who are undergoing angiography and stenting or surgery for treatment of their dissection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2005-11; Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor John W Norris, MD, FRCP, Principal Investigator — St George's, University of London; Professor Hugh Markus, DM, FRCP, Principal Investigator — St George's, University of London
Locations (1):
- St. George's University of London, Clinical Neuroscience Department, Cranmer Terrace, London, England, United Kingdom

REFERENCES:
- See also: Related Info — http://www.dissection.co.uk